CLINICAL TRIAL: NCT01748175
Title: Implications and Stability of Clinical and Molecular Phenotypes of Severe Asthma
Acronym: SARPIII
Status: Completed | Type: Observational
Sponsor: Sally E. Wenzel MD (Other)
Responsible Party: Sponsor-Investigator, Sally E. Wenzel MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: 1010HL109152-01
Record Dates: First submitted 2012-11-27; First posted 2012-12-12 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Asthma; Severe Persistent Asthma
Keywords: Severe asthma; longitudinal study; phenotypes
MeSH Terms: conditions — Asthma | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Longitudinal follow up: Patients will undergo a characterization phase, which includes a baseline evaluation (1 visit), and a steroid responsiveness evaluation (2 visits). The longitudinal phase will include 3 office visits (annually) over 36 months with bi-annual phone calls. During the study patients will answer questionnaires, perform lung function testing and provide blood, urine, sputum and exhaled breath condensate samples.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Each subject that meets inclusion/exclusion criteria will receive triamcinolone acetonide intramuscularly at the end of visit 2. Adults ≥18 years will receive 40 mg triamcinolone acetonide. Children 6-17 years will receive 1 mg/kg triamcinolone acetonide (up to 40 mg maximum). Triamcinolone acetonide will be administered as a single intramuscular dose deep in the gluteal region
  Other Names: Kenalog

SUMMARY:
The Severe Asthma Research Program III is an NIH cooperative agreement involving 7 clinical centers that encompass a multidisciplinary partnerships between asthma clinician-scientists and scientists with expertise in immunology, pulmonary physiology, molecular genetics, molecular phenotyping, imaging, and bioinformatics. These clinical centers will jointly recruit volunteers with asthma for an observational longitudinal follow-up study. However, centers will also conduct specific mechanistic research projects at each participating institution. The University of Pittsburgh's SARP III study will determine the molecular and clinical stability of asthma phenotypes over time.

DETAILED DESCRIPTION:
The longitudinal follow-up study is divided into a characterization and longitudinal phase. During the characterization subjects will undergo a baseline evaluation that will include will include answering questionnaires, lung function testing, and chest tomography. Subsequently, to determine steroid responsiveness, all subjects will receive one intramuscular dose of 40 mg in 1ml (1 mg/kg for children <18 years old, up to 40 mg maximum. Participants at the University of Pittsburgh will undergo a bronchoscopy to provide airway samples. The longitudinal phase will include a 36 month follow-up time with annual visits and phone calls every 6 months. During it, participants will answer questionnaires and provide sputum samples on two occasions, and will perform lung function testing.

The SARP III longitudinal follow up study (all centers) will determine the long term stability and implications of clinical and molecular asthma phenotypes and identify potential systemic biomarkers for these phenotypes

The University of Pittsburgh center will test the hypothesis that a) a mast cell signature is present and longitudinally maintained in severe asthma; and b) That the persistent signature determines short and long term outcomes through interactions with lung and inflammatory cells.

ELIGIBILITY:
Asthmatic Subjects

Inclusion Criteria:

* Previous asthma diagnosis
* FEV1 bronchodilator reversibility ≥12% or airway hyperresponsiveness reflected by a methacholine PC20 ≤16 mg/mL (Historical methacholine data from previous NIH trial [SARP I or II, AsthmaNet, ALA-ACRC, ACRN or CARE] will be allowed).

Exclusion Criteria:

* Exclusion criteria include any of the following:
* Pregnancy during the characterization phase
* Current smoking,
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age (Note: if a subject has a smoking history, no smoking within the past year),
* Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion), severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways,
* History of premature birth before 35 weeks gestation,
* Unwillingness to receive an intramuscular triamcinolone acetonide injection.
* Evidence that the participant or family may be unreliable or poorly adherent to their asthma treatment or study procedures,
* Planning to relocate from the clinical center area before study completion,
* Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician(s) of record, or
* Currently participating in an investigational drug trial.

Healthy Controls:

Inclusion Criteria

* Healthy subjects between the age of 18 and 65
* At least 3 of the 7 subjects per center should be aged 35 or older

Exclusion Criteria:

* History of chronic diseases that affect the lungs: Chronic airway disease (asthma, cystic fibrosis, COPD, chronic bronchitis, bronchiectasis); Interstitial lung disease, sarcoidosis, occupational lung disease; Obstructive sleep apnea; Vocal cord dysfunction; Severe scoliosis or chest wall deformities.
* A history suggestive of allergic rhinitis (based on the best judgment of the physician investigator).
* A history of eczema.
* Chronic sinusitis.
* An improvement in FEV1 of more than 12% following 4 puffs of albuterol.
* Chronic systemic diseases requiring ongoing anti-inflammatory treatment.
* Current use of beta adrenergic blocking agent or a cholinesterase inhibitor (medicine used to treat myasthenia gravis or Alzheimer's disease).
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age (Note: if a subject has a smoking history, no smoking within the past year).
* Respiratory tract infection within the past 4 weeks.
* Pregnancy.
* History of premature birth (<35 weeks).
* Any other criteria that place the subject at increased risk of complications from study procedures, according to the judgment of the Principal Investigator and/or attending physician(s) of record.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with asthma meeting inclusion and exclusion criteria will be recruited from 7 SARP III participating clinical centers. The clinical centers are located at Brigham and Women's Hospital (with co-investigators at Children's Hospital), the University of California San Francisco, the University of Pittsburgh, the University of Virginia (with co-investigators at the Cleveland Clinic, Case Western Reserve and Virginia Commonwealth University), the University of Wisconsin, Wake Forest School of Medicine (with co-investigators at Emory University), and Washington University in St. Louis (with co-investigators at the University of Iowa).
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2013-01; Primary Completion 2021-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Airway lumen mast cells | Once, during bronchoscopy
  Determine the impact of mast cell markers on human airway epithelial cell phenotype and function.
Longitudinal asthma phenotype | Change rates, determined annually for three years
  Determine the long term stability and implications of previously identified clinical and molecular asthma phenotypes, specifically the mast cell signature, and identify potential systemic biomarkers for these phenotypes.
  Determine whether a biomarker for the lung mast cell signature can be identified in serum/plasma of both adult and pediatric severe asthmatics

CONTACTS AND LOCATIONS:
Overall Officials: Sally E Wenzel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Asthma Institute, UNiversity of Pittsburgh and University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] DeBoer MD, Phillips BR, Mauger DT, Zein J, Erzurum SC, Fitzpatrick AM, Gaston BM, Myers R, Ross KR, Chmiel J, Lee MJ, Fahy JV, Peters M, Ly NP, Wenzel SE, Fajt ML, Holguin F, Moore WC, Peters SP, Meyers D, Bleecker ER, Castro M, Coverstone AM, Bacharier LB, Jarjour NN, Sorkness RL, Ramratnam S, Irani AM, Israel E, Levy B, Phipatanakul W, Gaffin JM, Gerald Teague W. Effects of endogenous sex hormones on lung function and symptom control in adolescents with asthma. BMC Pulm Med. 2018 Apr 10;18(1):58. doi: 10.1186/s12890-018-0612-x. PMID 29631584

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT01748175/Prot_SAP_000.pdf